CLINICAL TRIAL: NCT04387110
Title: Monoclonal Antibodies in Mothers' Milk and Infants: Ocrelizumab in Breastmilk
Brief Title: Ocrelizumab in Breastmilk
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-22422
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breastmilk-Breastmilk will be serially sampled prior to and after the first infusion(s) postpartum according to the following schedule:
  * 600mg infusion x1: before infusion and at 8H, 24H, 7D, 20D, 30D, 60D, and 90D post
  * 300mg infusion x2: before infusion 1, at 8H, 24H, 7D, and 14D (before infusion 2) after infusion 1 and after infusion 2 at 8H, 24H, 7D, 20D, 30D, 60D, and 90D
  Blood (serum)- Samples will be collected to determine maternal serum concentration of ocrelizumab relative to breastmilk samples at the following timepoints:
  * 600mg infusion x1: 24H and 20D post infusion
  * 300mg infusion x2: 24H and 14D (post infusion 1) and 24H and 20D (post infusion 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Ocrelizumab: Women receiving treatment for multiple sclerosis with ocrelizumab infusion between 2 and 36 weeks postpartum.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Receiving either 1infusion (600mg) or 2 infusions (300mg).
  Other Names: ocrevus

SUMMARY:
The goal of the current project is to measure the levels of ocrelizumab in the breastmilk of women with multiple sclerosis (MS) and clinically isolated syndrome (CIS) who are postpartum, and to collect information on 12-month infant development outcomes (length, weight, head circumference, infections) in their offspring.

This study will fill a significant unmet need as many women with MS at high risk for postpartum relapses are not effectively treated for their MS in the postpartum period due to lack of information about the presence, concentration and effects of medications in breastmilk.

DETAILED DESCRIPTION:
Levels of ocrelizumab in breastmilk will be serially evaluated across one drug half-life from women with MS and CIS who are postpartum and lactating at the time of the infusion (whether or not they plan to continue to breastfeed their baby after the infusion). The timeline for breastmilk sample is dependent on infusion schedule and dosing if receiving 600mg infusion x1, collection will occur: before infusion and at 8H, 24H, 7D, 20D, 30D, 60D, and 90D post infusion; if receiving 300mg infusion x2 collection will occur: before infusion 1, at 8H, 24H, 7D, and 14D (before infusion 2) after infusion 1 and after infusion 2 at 8H, 24H, 7D, 20D, 30D, 60D, and 90D in 20. Blood samples to determine serum concentration of ocrelizumab will be collected, when possible, at the 24-hour, 14 day (if receiving 300mg infusion x2), and 20D timepoint(s). Both women continuing to breastfeed their infant post-infusion and those that chose to discontinue will be included in the study.

In order to ensure broad collaboration as well as rapid recruitment, samples will be collected from patients fitting eligibility criteria upon referral to our study by other investigators.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 64 that carry a diagnosis of Clinically Isolated Syndrome or Multiple Sclerosis (based on the 2010 McDonald Criteria).
* Participants must be pregnant, contemplating pregnancy or postpartum at the time of enrollment.
* Participants must be receiving treatment with ocrelizumab infusion between 2 and 36 weeks postpartum (300mg x2 or 600mg x1).
* Participants must be willing to provide breastmilk samples before and after their first and, if applicable, second ocrelizumab infusions postpartum.
* A signed informed consent and HIPAA authorization form is required for participation.

Exclusion Criteria:

* Patients unable to provide informed consent.
* Patients unable or unwilling to provide breast milk samples for analysis.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Study participants will be identified via self referral from study advertisements (via the National MS Society and clinicaltrials.gov) or referred by clinician at the UCSF MS Center.
  Clinicians outside of UCSF will also be invited to refer eligible patients to the study by providing study team contact information.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Determine levels of ocrelizumab in the breastmilk of women with MS | 12 months
  Levels of ocrelizumab (μg/mL) in the breastmilk of women at the selected timepoints before and after infusion (hour 8, hour 24, day 7, day 20, day 30, day 60, and day 90). If receiving two infusions the samples will be as follows: pre-infusion, hour 8, hour 24, day 7, and day 14 after infusion 1(prior to infusion 2); then post infusion 2, at hour 8, hour 24, day 7, day 20, day 30, day 60, and day 90. This outcome will be measured by breastmilk concentration (μg/mL), average breastmilk concentration (CAVE, determined using pharmacokinetic methods), maximum concentration of ocrelizumab in breastmilk (CMAX), absolute average ocrelizumab dose to the infant in a 24-hour period, maximum ocrelizumab dose to the infant in a 24-hour period, average relative infant dose (RIDAVE), and maximum relative infant dose (RIDMAX).
Determine time to peak levels of ocrelizumab in the breastmilk of women with MS. | 12 months
  Based on analysis of levels of ocrelizumab (μg/mL) in the breastmilk of women at the selected timepoints before and after infusion (hour 8, hour 24, day 7, day 20, day 30, day 60, and day 90). If receiving two infusions the samples will be as follows: pre-infusion, hour 8, hour 24, day 7, and day 14 after infusion 1(prior to infusion 2); then post infusion 2, at hour 8, hour 24, day 7, day 20, day 30, day 60, and day 90. The average peak level of ocrelizumab concentration will be determined.
Determine predictors of ocrelizumab levels in breastmilk. | 12 months
  The following predictors will be assessed in relation to level of detectable ocrelizumab in breastmilk: ocrelizumab dosing (300 vs. 600mg), maternal age and parity, introduction of solid foods, and other clinical factors.

SECONDARY OUTCOMES:
Obtain information on newborn adjusted length until 12 months of life. | 12 months
  Newborn adjusted length (in cm) will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn weight until 12 months of life. | 12 Months
  Newborn weight (in kg) will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn head circumference until 12 months of life. | 12 Months
  Newborn head circumference (in cm) will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn infections until 12 months of life. | 12 Months
  Newborn infections will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn vaccines until 12 months of life. | 12 Months
  Newborn vaccine completed and scheduled vaccines will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn developmental milestones until 12 months of life. | 12 Months
  The Ages and Stages Questionnaire, third edition, (ASQ-3) will be completed by participating mothers at the following timepoints postpartum, to determine the developmental age of infants: 2 months, 4 months, 6 months, 8 months, 10 months and 12 months. The questionnaire scores 5 areas of development: Communication, Gross Motor, Fine Motor, Problem Solving and Personal-Social. Cumulative scores range from 0 to 60. Higher scores indicate more positive outcomes. Each version of the ASQ-3 has different cutoff scores that indicate whether the child's development appears to be on schedule, requires monitoring or requires further assessment. (Above and Monitoring Ranges indicate on schedule infant development for age).

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genentech. (2011). Prescribing Information. [PDF File]. Retrieved from https://www.gene.com/download/pdf/ocrevus_prescribing.pdf
- [Background] Matro R, Martin CF, Wolf D, Shah SA, Mahadevan U. Exposure Concentrations of Infants Breastfed by Women Receiving Biologic Therapies for Inflammatory Bowel Diseases and Effects of Breastfeeding on Infections and Development. Gastroenterology. 2018 Sep;155(3):696-704. doi: 10.1053/j.gastro.2018.05.040. Epub 2018 May 30. PMID 29857090
- [Background] Hale TW, Rowe HE. Medications and mothers' milk. 16th ed. Amarillo (TX): Hale Publishing; 2014
- [Background] Krysko KM, LaHue SC, Anderson A, Rutatangwa A, Rowles W, Schubert RD, Marcus J, Riley CS, Bevan C, Hale TW, Bove R. Minimal breast milk transfer of rituximab, a monoclonal antibody used in neurological conditions. Neurol Neuroimmunol Neuroinflamm. 2019 Nov 12;7(1):e637. doi: 10.1212/NXI.0000000000000637. Print 2020 Jan. PMID 31719115